CLINICAL TRIAL: NCT01971047
Title: The Safety and Efficacy of Correcting Preoperative Hyperglycemia in Ambulatory Surgical Patients With Diabetes: A Randomized Controlled Clinical Trial
Brief Title: Safety and Efficacy Study of Correcting Hyperglycemia in Patients With Diabetes Having Out-patient Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Karen Carlson, MD, Study Principal Investigator, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00067662
Record Dates: First submitted 2013-09-26; First posted 2013-10-28 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-03

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
Keywords: Diabetes; Surgery; anesthesiology; endocrinology
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Insulin; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1-Regular Insulin (Active Comparator): Intravenous Regular Insulin will be administered for a preoperative Blood glucose of greater than 180.
  Interventions: Drug: Regular Insulin
- Group 2-Humalog (Active Comparator): Subcutaneous Humalog will be administered for a preoperative Blood glucose of greater than 180
  Interventions: Drug: Humalog

INTERVENTIONS:
Drug: Regular Insulin — Group 1 Treatment Arm,Follow dosing for BG >180 per the following formula:
  1. Patients with Type 2 Diabetes to receive dosage based on the formula: (BG-120)/30= # units of insulin
  2. Patients with Type 1 Diabetes to receive dosage based on the formula: (BG-120)/40=# units of insulin
  3. Patients with Type 1 Diabetes and Type 2 Diabetes over the age of 70 or with chronic kidney disease to receive dosage based on the formula: (BG-120)/50=# units of insulin
  4. Consider repeating dose if BG>240 mg/dl after 2 hours of initial dose
  Other Names: Novolin
  Arms: Group 1-Regular Insulin
Drug: Humalog — Group 2 treatment arm. Follow dosing for Blood glucose > 180, per the following formula:
  1. Patients with Type 2 Diabetes to receive dosage based on the formula: (BG-120)/30= # units of insulin
  2. Patients with Type 1 Diabetes to receive dosage based on the formula: (BG-120)/40=# units of insulin
  3. Patients with Type 1 Diabetes and Type 2 Diabetes over the age of 70 or with chronic kidney disease to receive dosage based on the formula: (BG-120)/50=# units of insulin
  4. Consider repeating dose if BG>240 mg/dl after 2 hours of initial dose
  Other Names: Lispro
  Arms: Group 2-Humalog

SUMMARY:
The purpose of this study is to compare the safety and efficacy of intravenous (IV) administration of FDA approved regular human insulin and subcutaneous (SC) administration of humalog, a rapid-acting insulin analog (a synthetic insulin), for correction of hyperglycemia (high blood sugar) during the immediate preoperative period in patients with diabetes having outpatient surgery at the Emory Ambulatory Surgical Center (ASC).

In this randomized controlled clinical trial patients with diabetes will be administered corrective doses of IV regular insulin or SC humalog for preoperative hyperglycemia to determine whether SC humalog results in improved intra and post-operative blood sugar control.The most common current practice at Emory University in the ambulatory surgical setting is IV administration of regular insulin for treatment of pre-operative hyperglycemia. Subjects will not be paid for their participation and will be assured of treatment for their hyperglycemia regardless of study participation.

DETAILED DESCRIPTION:
Investigators plan to randomize a total of 200 male and female subjects with type 1 and type 2 diabetes,having an out patient surgical procedure, meeting inclusion criteria to receive corrective doses of IV regular insulin (Group I) or SC humalog insulin (Group II). The dosing formula is per Emory University Outpatient Surgical Center protocol for treating hyperglycemia and is the same for both groups. All patients with diabetes will undergo a blood sugar measurement upon arrival to the ASC using the Accuchek blood glucose meter. An admission blood sugar of >180 in a patient with diabetes qualifies the patient for study screening. Subjects will be approached after confirmation of eligibility for the study. Randomization, then treatment, will occur immediately following written informed consent. Demographic data will be recorded.A medical history with detailed history of diabetes will be obtained and surgical and anesthesia details and length of stay recorded. Blood sugar levels will be checked hourly until the patient is ready for discharge. Subsequent treatment will follow the hyperglycemia protocol. All blood sugar results and doses of insulin will be recorded. The subject's participation will end at the time of discharge from the Ambulatory Surgical Center.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 80 years with type 1 and type 2 diabetes
* patients undergoing ambulatory surgery
* a known history of diabetes for > 3 months treated with diet, oral antidiabetic agents and/or insulin therapy
* subjects with an admission/randomization Blood glucose> 180 and < 400 mg/dl
* Patients willing and able to provide informed consent

Exclusion Criteria:

* Age < 18 or > 80
* Subjects with increased blood glucose concentration, but without a history of diabetes (stress hyperglycemia)
* Patients on an insulin pump
* Patients with a history of clinically significant hepatic disease (cirrhosis, jaundice, end-stage liver disease, portal hypertension) and end- stage renal disease
* Current or recent (within 3 months) treatment with oral or injectable corticosteroid, parenteral nutrition and immunosuppressive treatment
* Mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study
* Female subjects whom are pregnant or breast-feeding at time of qualifying outpatient procedure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
BG concentration differences at 1 and 2 hours post intervention and post operatively | one and two hours post intervention, post operative period
  Compare the difference in Blood glucose concentration at one and two hours after the administration of corrective doses of regular and humalog insulin and immediately following ambulatory surgery.

SECONDARY OUTCOMES:
Number and percentage of target BG readings | From time of treatment until patient discharge (an average of three hours, less than one day)
  Investigators will determine the number and percentage of patients in each group with BG readings within the target range ( 80-180 mg/dl)
Episodes of hypoglycemia | time of intervention to time of patient discharge (an average of three hours, less than one day)
  Investigators will assess if there is any difference in the number of hypoglycemic events between the two treatment groups and further assess the rate and frequency of hypoglycemia (<70 mg/dl) and severe hypoglycemia (<40 mg/dl).
Episodes of hyperglycemia | time of treatment to time of patient discharge (an average of three hours, less than one day)
  Investigators will calculate the number of patients and percent of BG readings with hyperglycemia (>180 mg/dl) and severe hyperglycemia (>300 mg/dl)in each group.
Total dose of insulin | time of intervention to time of patient discharge (an average of three hours, less than one day)
  Calculate total dosage of insulin administered to each patient
Change in glucose concentration from baseline to one, two and three hours post treatment | time of baseline BG to time of last BG measurement (prior to discharge, less than one day)
  Change in glucose concentration from baseline (prior to insulin administration) to one hour, two hours and three hours (if patient present) after insulin administration
Number of perioperative complications | start of surgery to time of patient discharge (less than one day)
  Investigators will record the number of perioperative complications (cardiovascular, respiratory or other medical complications) or need for hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Carlson Karen, MD, Principal Investigator — Emory University
Locations (1):
- Emory Healthcare Ambulatory Surgical Center, Atlanta, Georgia, United States